CLINICAL TRIAL: NCT02461446
Title: Natural History Study of Individuals With Autism and Germline Heterozygous PTEN Mutations
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mustafa Sahin, Professor of Neurology, Harvard Medical School, Boston Children's Hospital
Other Study IDs: P00013150; 1U54NS092090-01 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2015-06-03 (Estimated); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: PTEN; ASD; Autism; Macrocephaly; PTEN Hamartoma Tumor Syndrome
Keywords: germline heterozygous PTEN mutations; MRI; 10q23.3; ASD; Autism; Macrocephaly; PTEN Hamartoma Tumor Syndrome; PTEN; EEG
MeSH Terms: conditions — Autistic Disorder; Megalencephaly; Hamartoma Syndrome, Multiple

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draw for future correlative studies in the PTEN Biorepository of the Developmental Synaptopathies Consortium.
  170 subjects; 100 existing subjects, 70 newly enrolled participants; 50 controls
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PTEN ASD: PTEN participants with Autism Spectrum Disorder group
- PTEN no ASD: PTEN participants without Autism Spectrum Disorder group
- Controls: Healthy control group

SUMMARY:
The purpose of this study is to determine cross-sectional and longitudinal medical, behavioral, and cognitive differences between PTEN ASD and other groups, as well as to identify cognitive, neural systems, and molecular biomarkers specific to PTEN ASD. In addition, this study will be creating and maintaining a biorepository and linked phenotypic database for PTEN ASD.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) are a set of neurodevelopmental disorders characterized by social communication/interaction impairments and restricted/repetitive behaviors. ASD associated with germline heterozygous PTEN mutations (PTEN ASD) is a genetically defined sub-group that, may be one of the more prevalent genetic disorders contributing to ASD (0.5-2%). The purpose of this research study is to carefully track the phenotypic and molecular characteristics of PTEN ASD and identify biomarkers for intervention studies.

Individuals with PTEN ASD, with macrocephalic ASD without a PTEN mutation (macro-ASD), healthy controls, and individuals with PTEN mutations without ASD (PTEN no-ASD) will be asked to participate in this study if they are 18 months and older. Both males and females will be asked to participate. Additionally, to be eligible for study participation, individuals' primary communicative language must be English.

The study involves 3 on site visits over the course of two years. Study visits will vary in length from about 4 hours to 6 hours. Study visits involve a physical exam, medical history questions, neuropsychological assessments, and a blood draw done for laboratory studies. A subset of participants between the ages of 2 and 11 years old will take part in the EEG portion of the study. Individuals who have a clinically indicated MRI will have an option to provide routine clinical scans for analysis.

ELIGIBILITY:
Inclusion Criteria

* Individuals above the age of 18 months old at the time of consent who have documentation of a clinical diagnosis of autism spectrum disorder and/or a verified PTEN mutation from a medical or mental health professional for inclusion in the PTEN ASD, PTEN no-ASD or ASD macrocephaly groups.
* Macrocephaly (head circumference greater than or equal to 98th percentile) for inclusion in the ASD macrocephaly group.
* For youths, consent from parents or legal guardian. For adults, consent from self or legal guardian.
* Youths who are able (some young or severely impaired participants may not be able to provide assent) will be asked to provide assent as per IRB guidelines.
* Families with multiple children who meet the above inclusion criteria will be permitted to have as many children participate as they wish. A separate consent form will be filled out for each child enrolled in the study.
* Primary communicative language must be English

Exclusion Criteria

* Unwilling or unable to comply with study procedures and assessments
* Clinically significant medical disease that would prohibit participation in the study procedures.
* For subjects ELIGIBLE FOR OPTIONAL imaging biomarker assessment: contraindications to 3T MRI scanning, such as metal implants/non-compatible medical devices or medical conditions, including vagus nerve stimulator.
* For subjects ELIGIBLE FOR EEG/ERP biomarker assessment: contraindications to EEG/ERP, such as uncooperative or destructive behaviors preventing lead placement or capture by ERP/VEP equipment. Under age 2 or over 11 at the time of enrollment.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 170 patients will be enrolled for this study, over the age of 18 month old.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2015-05; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in verbal abilities at 12 months | 12 months
  Verbal and non-verbal ability will be evaluated using Stanford Binet -5 or Mullen Scales of Early Learning (MSEL) at 12 months
Change in communication ability at 12 months | 12 months
  Communication ability will be evaluated using composite score of the Peabody Picture Vocabulary Test (PPVT-4).
Change in communication ability at 12 months | 12 months
  Communication ability will be evaluated using composite score of the Expressive Vocabulary Test (EVT-2) at 12 months.
Change in verbal abilities at 24 months | 24 months
  Verbal and non-verbal ability will be evaluated using Stanford Binet 5 or Mullen Scales of Early Learning (MSEL) at 24 months
Change in visual perception at 12 months | 12 months
  Visual perception will be measured using the Beery Developmental Test of Visuomotor Integration (VMI) at 12 months
Change in working memory at 12 months | 12 months
  Working memory will be evaluated using the Stanford Binet 5 at 12 months
Change in processing speed at 12 months | 12 months
  Processing Speed will be measured using the Processing Speed Index from the Weschler Intelligence Scales at 12 months
Change in working memory at 24 months | 24 months
  Working memory will be evaluated using the Stanford Binet 5 at 24 months
Change in processing speed at 24 months | 24 months
  Processing Speed will be measured using the Processing Speed Index from the Weschler Intelligence Scales at 24 months
Change in visual perception at 24 months | 24 months
  Visual perception will be measured using the Beery Developmental Test of Visuomotor Integration (VMI) at 24 months
Change in communication ability at 24 months | 24 months
  Communication ability will be evaluated using composite score of the Peabody Picture Vocabulary Test (PPVT-4) at 24 months
Change in communication ability at 24 months | 24 months
  Communication ability will be evaluated using composite score of the Expressive Vocabulary Test (EVT-2) at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hardan, MD, Study Chair — Stanford University
Locations (5):
- United States (5):
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Frazier TW, Jaini R, Busch RM, Wolf M, Sadler T, Klaas P, Hardan AY, Martinez-Agosto JA, Sahin M, Eng C; Developmental Synaptopathies Consortium. Cross-level analysis of molecular and neurobehavioral function in a prospective series of patients with germline heterozygous PTEN mutations with and without autism. Mol Autism. 2021 Jan 28;12(1):5. doi: 10.1186/s13229-020-00406-6. PMID 33509259